CLINICAL TRIAL: NCT00193674
Title: Oral Dydrogesterone Treatment During the First Trimester of Pregnancy in Women With Recurrent Miscarriage: A Double-Blind, Prospectively Randomized, Placebo-Controlled, Parallel Group Trial
Brief Title: Habitual Abortion Study: Oral Dydrogesterone Treatment During Pregnancy in Women With Recurrent Miscarriage
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Products (Industry)
Responsible Party: Sponsor
Organization: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S102.3.116
Record Dates: First submitted 2005-09-11; First posted 2005-09-19 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2011-08

CONDITIONS: Recurrent Miscarriage
Keywords: Pregnancy; Immunology; Unexplained recurrent miscarriage
MeSH Terms: conditions — Abortion, Habitual | interventions — Dydrogesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Dydrogesterone
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dydrogesterone — 20 mg/day, oral
  Arms: 1
Drug: Placebo — Placebo
  Arms: 2

SUMMARY:
The purpose of this clinical study is to demonstrate the shift from inflammatory cytokines to non-inflammatory cytokines in women suffering from habitual abortion treated with dydrogesterone (Duphaston).

ELIGIBILITY:
Inclusion Criteria

* Women with a history of idiopathic recurrent miscarriage, based on a documented history of at least three spontaneous consecutive miscarriages before 20 weeks gestation with the same partner Exclusion Criteria
* Any verifiable cause of the recurrent miscarriages apart from luteal phase defect (e.g. systemic lupus erythematosus [SLE], infections with chlamydia or mycoplasma)
* Any gynecological neoplasias or anatomical abnormalities that oppose pregnancy
* Concurrent infertility treatment/superovulation protocol

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2003-09; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Cytokine ratio IFN/IL-10 | 14 weeks treatment after diagnosed pregnancy (week of gestation 4 to 18)

SECONDARY OUTCOMES:
Exploratory analysis of pregnancy outcome by monitoring biochemical and clinical pregnancy parameters, weekly evaluation of serum progesterone | First trimester of pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Guenter Krause, MD, Study Director — Abbott Products
Locations (3):
- Site Reference ID/Investigator# 61182, Vienna, Austria
- Poland (2):
  - Site Reference ID/Investigator# 61183, Poznan
  - Site Reference ID/Investigator# 61184, Szczecin